CLINICAL TRIAL: NCT05328752
Title: A Randomized, Participant- and Investigator-blinded, Sponsor Open-label, Placebo-controlled, Single and Multiple Dose Study to Investigate the Safety and Tolerability of XXB750 in Heart Failure Participants With Reduced or Mildly Reduced Ejection Fraction (HFrEF/HFmrEF)
Brief Title: Safety and Tolerability Study of XXB750 in Heart Failure Participants With Reduced or Mildly Reduced Ejection Fraction (HFrEF/HFmrEF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXXB750A12101; 2021-006683-24 (EudraCT Number)
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); or Heart Failure With Mildly Reduced Ejection Fraction (HFmrEF)
Keywords: heart failure; reduced ejection fraction; mildly reduced ejection fraction; HFrEF; HFmrEF; XXB750
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled safety study of XXB750
Who Masked: Participant, Care Provider
Masking Description: Site will have masked and unmasked investigators. An unmasked investigator will prepare and administer dose while a masked investigator will perform all assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- XXB750 Cohort 1 (Experimental): XXB750, single dose
  Interventions: Drug: XXB750
- Placebo Cohort 1 (Placebo Comparator): Placebo, single dose
  Interventions: Drug: Placebo
- XXB750 Cohort 2 (Experimental): XXB750, multiple doses
  Interventions: Drug: XXB750
- Placebo Cohort 2 (Placebo Comparator): Placebo, multiple doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XXB750 — XXB750
  Arms: XXB750 Cohort 1; XXB750 Cohort 2
Drug: Placebo — Placebo
  Arms: Placebo Cohort 1; Placebo Cohort 2

SUMMARY:
This is a multi-center, randomized, sponsor open-label, participant- and investigator-blinded, placebo-controlled, single and multiple dose study to investigate the safety and tolerability of XXB750 in HFrEF/HFmrEF.

DETAILED DESCRIPTION:
A screening period of up to 29 days will be used to assess participants' eligibility. This study will consist of 2 cohorts. Cohort 1 will include participants on stable therapies of ACEi/ARB and beta-blockers, in addition to other standard of care medications. Cohort 2 will consist of participants treated with sacubitril/valsartan and beta-blockers, in addition to other standard of care medications.

For Cohort 1 participants will be randomized in a 2:1 ratio to receive a single dose of subcutaneous (s.c) XXB750 or placebo. For Cohort 2, participants will be randomized in a 3:1 ratio to receive three doses of either s.c. XXB750 or placebo.

Cohort 1: After an initial domiciling period following study drug administration, participants will be followed for 13 weeks post-dosing for safety, tolerability and PK until the End of Study visit on Day 91.

Cohort 2: After a domiciling period following first study drug administration of XXB750 or placebo, participants will be followed for 27 days post dosing for safety, tolerability and PK. On Day 28, participants will be re domiciled and receive a second dose of either XXB750 or placebo. Participants will be followed for another 27 days post-dosing for safety and tolerability. On Day 56, participants will be re-domiciled and receive a third dose of either XXB750 or placebo. After the third domiciling period, participants will be followed for 13 weeks post-dosing for safety, tolerability and PK until the End of Study visit on Day 146.

ELIGIBILITY:
Key Inclusion Criteria:

* NYHA functional class II-III
* LVEF ≤ 50% documented at screening
* Systolic blood pressure 110 - 160 mmHg (cohort 1) or 105-160 mmHg (cohort 2), and heart rate between 50-90 beats per minute, inclusive
* Treatment with a stable dose of a beta blocker.
* Cohort 1: Treatment with a stable dose of ACE inhibitor or ARB
* Cohort 2: Treatment with a stable dose of sacubitril/valsartan.

Key Exclusion Criteria

* Acute decompensated heart failure within 3 months prior to screening. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid, or other major cardiovascular surgery, PCI, or carotid angioplasty within the 6 months prior to screening
* Hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to LV dilatation at screening
* Implantation of a CRT device within 3 months prior to screening or intent to implant a CRT during the study period
* History of severe pulmonary disease (e.g. COPD) requiring chronic supplemental oxygen therapy or pulmonary hypertension requiring pharmacology treatment at Screening
* eGFR <45 mL/min/1.73 m2 at screening
* Cohort 1 only: Treatment with sacubitril/valsartan currently or within 4 weeks from screening
* Cohort 2: Treatment with ACE inhibitor or ARB currently or within 4 weeks from screening
* BMI >40 kg/m2

Other protocol-specific criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Adverse events, which may include abnormal vital signs, safety lab tests, or ECG parameters that induce clinical signs or symptoms, are considered clinically significant or require therapy | 91 days (Cohort 1), 146 days (Cohort 2)
  To evaluate the safety and tolerability of XXB750 in adult participants with chronic stable heart failure with reduced or mildly reduced ejection fraction (HFrEF/HFmrEF).

SECONDARY OUTCOMES:
Pharmacokinetics parameters Tmax | 91 days (Cohort 1), 146 days (Cohort 2)
  To evaluate the pharmacokinetics: Time to maximum concentation (Tmax) parameters of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters Cmax | 91 days (Cohort 1), 146 days (Cohort 2)
  To evaluate the pharmacokinetics parameters: Peak plasma concentration (Cmax) of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters AUClast for Cohort 1 | 91 days
  To evaluate the pharmacokinetics parameters: Area under the plasma concentration curve (AUClast) of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters AUCinf for Cohort 1 | 91 days
  To evaluate the pharmacokinetics parameters: Area under the curve (AUCinf) of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters Vz/F | 91 days (Cohort 1), 146 days (Cohort 2)
  To evaluate the pharmacokinetics parameters: Vd/F of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters CL/F | 91 days (Cohort 1), 146 days (Cohort 2)
  To evaluate the pharmacokinetics parameters: (CL/F) of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters T1/2 | 91 days (Cohort 1), 146 days (Cohort 2)
  To evaluate the pharmacokinetics parameters: (T1/2) of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.
Pharmacokinetics parameters AUCtau for Cohort 2 | 146 days
  To evaluate the pharmacokinetics parameters: Area under the curve (AUCtau) of XXB750 in adult participants with chronic stable HFrEF/HFmrEF.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (3):
  - Nature Coast Clinical Research LLC, Inverness, Florida
  - Jacksonville Ctr for Clin Rea Main Centre, Jacksonville, Florida
  - Fairview Health Services ., Saint Paul, Minnesota
- Novartis Investigative Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CXXB750A12101 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18250
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2455